CLINICAL TRIAL: NCT04796883
Title: A Study for Assessing the Safety of Hanita Glaucoma Shunt in Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGS-01
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Hanita Glaucoma shunt Ver.3.2
  Interventions: Device: Hanita Glaucoma shunt Ver.3.2

INTERVENTIONS:
Device: Hanita Glaucoma shunt Ver.3.2 — The procedure will be performed under anesthesia (at physician discretion) and a Hanita shunt devce will be implanted.

SUMMARY:
The HANITA Glaucoma Filtration Device is intended to reduce intraocular pressure in glaucoma patients where medical and conventional surgical treatments have failed.

DETAILED DESCRIPTION:
Study Design:

This study is a prospective, single-arm single-center, open-label study.

Study population:

Men and women diagnosed with open-angle glaucoma who require glaucoma surgery procedures that meet the inclusion/exclusion criteria and provide written informed consent will be enrolled in the study.

Enrollment:

A total of 30 subjects will be enrolled:

15 patients will be implanted according to procedure 1 (see section 8.7), at completion additional 15 patients will be implanted according to procedure 2 (see section 8.7)

Investigational sites:

One (1) center will participate in this study.

Duration of Subject participation:

Completion of active enrolment is anticipated to last approximately 6 months. The primary endpoint will be achieved when the final study subject has completed 6 months follow-up.

Study Group:

A single study group. This is a single-arm design; there is no control device in this study.

Visits & Procedures Pre-operative visit: 0-3 months prior to the implantation procedure. The visit will include the subject's qualification assessment for inclusion/exclusion criteria as described above. Informed consent must be signed.

Complete anamnesis will be taken including the subject's medical complaints, medical history, and medication use. Ophthalmic examinations as well as ultrasound biomicroscopy.

Surgical procedure: Procedure will be performed under anesthesia (at physician discretion) and a Hanita shunt will be implanted.

Follow-up: All subjects will have regular follow-up visits at 1 and 7 days and on 1, 3, and 6 months post-implantation. 1-year post-operative evaluation is optional at the sponsor's discretion. All postoperative visits will include a complete ophthalmic examination,

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 40 and 80 years of age
* Subject diagnosed with primary Open-angle glaucoma
* Subject is Diagnosed with glaucoma uncontrolled by medical therapy which meets at least one of the following criteria:
* Failed one or more incisional intraocular glaucoma surgeries (e.g., glaucoma filtering surgery or tube shunt)
* Failed one or more cilioablative procedures (e.g., cryotherapy, cyclodiode therapy)
* Have any other condition (e.g., conjunctival scarring, uveitis) in which a conventional incisional glaucoma surgery like trabeculectomy would be more likely to fail than for a person with uncomplicated primary open-angle glaucoma
* Under present-day criteria subject is a candidate for glaucoma surgery
* Intraocular pressures of the eye above or equal to 25 mmHg with or without medication
* The angle should be grade 3 in at least the 180º superior and not less than grade 2 at any level of the angle
* Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed

Exclusion Criteria:

* Subject diagnosed with primary angle-closure glaucoma (PACG)
* Subject diagnosed with normal-tension glaucoma (NTG)
* Subject diagnosed with secondary glaucoma
* Subject diagnosed with neovascular glaucoma
* Patient eyes with no light perception vision
* Patient eyes with the need for a combined glaucoma procedure or anticipated need for additional ocular surgery or retinal laser procedure within the 6-month follow-up period
* Patient eyes that have failed laser trabeculoplasty but have not met the stated inclusion criteria
* The subject has best-corrected visual acuity (BCVA) worse than 20/200 in the non-study eye
* Subject consumes the anti aggregating or anticoagulant and cannot suspend the use at least four days prior to the procedure, and antiplatelet drugs one week before
* The subject is diagnosed with glaucoma-related to other comorbidities (especially neovascular glaucoma, inflammatory glaucomas, glaucomas associated with hemorrhages and pseudoexfoliation)
* Subject with inadequate space in the anterior chamber and/or angle as determined by slit-lamp examination and gonioscopy
* The subject is diagnosed with active anterior segment intraocular inflammation
* The subject is obligated to previous participation in another study with any investigational drug or device within the past 30 days
* Subject is pregnant

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
VISUAL ACUITY | 1 year
  • Distance (far) manifest refraction and the testing distance used will be recorded on the case report forms. Manifest refraction will be determined using the maximum plus for best visual acuity method. The distance manifest refraction will be done with a distance adjusted chart but not less than 4 meters. The actual manifest refraction distance will be noted on the case report forms.
  Visual acuity will be measured with ETDRS format charts for distance and near. Results will be recorded in a LogMar scale.
SLIT LAMP EXAM | 1 year
  The slit lamp exam will include the measurement of aqueous cell and flare, and the measurement of corneal edema by a standard grading system. It will also include an evaluation for the presence of pupillary irregularities, iris atrophy and pigment dispersion. A gonioscopic exam using a consistent grading system at each site will also be conducted.
  For the evaluation of aqueous cells and flare, use a slit lamp beam 0.3 mm wide and 1 mm high, and use the following grading:
  Cells none (0) = no cells seen trace (+1) = 1-5 cells seen mild (+2) = 6-15 cells seen moderate (+3) = 16-30 cells seen severe (+4) = > 30 cells seen
  Flare none (0) = No Tyndall effect trace (+1) = Tyndall effect barely discernible mild (+2) = Tyndall beam in anterior chamber is mildly intense moderate (+3) = Tyndall beam in anterior chamber is moderately intense severe (+4) = Tyndall beam is severely intense. The aqueous has a white and milky appearance.
MEASUREMENT OF INTRAOCULAR PRESSURE | 1 year
  Intraocular pressure will be measured using Goldmann applanation tonometry or other validated methods.

CONTACTS AND LOCATIONS:
Locations (1):
- VISSUM, Madrid, Spain